CLINICAL TRIAL: NCT05760118
Title: Awareness of Osteoporosis in Diabetes Mellitus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: OPDM1
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Osteoporosis; Osteoporosis Risk
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetes Mellitus Patients: Patients diagnosed with diabetes mellitus.
  Interventions: Other: Patient Participation Form

INTERVENTIONS:
Other: Patient Participation Form — A form that consists of revised osteoporosis knowledge test, osteoporosis self-efficacy scale, and osteoporosis health belief scale.

SUMMARY:
Osteoporosis is a condition that describes compromised skeletal microarchitecture in general, with clinical signs of decreased bone mineral density. Diabetes mellitus patients are at increased risk for developing osteoporosis. Identifying whether multiple sclerosis patients have information and awareness about this disease is crucial. This study is aimed to investigate awareness and knowledge of osteoporosis in diabetes mellitus patients.

DETAILED DESCRIPTION:
Osteoporosis is a common disease of bone loss. The reduced bone strength predisposes an increased risk for fractures in older individuals. It can affect people from different ethnicity. Many factors increase the risk of osteoporosis, including age, postmenopausal state, glucocorticoid use, low body weight, calcium, vitamin D, immobility, and chronic inflammation. Patients with multiple sclerosis are at high risk of developing osteoporosis due to chronic inflammation and their medications. Patients' knowledge and awareness about osteoporosis are essential for early detection, implementation of lifestyle changes, and treatment compliance. This study aimed to investigate osteoporosis awareness and knowledge about osteoporosis in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes mellitus
* Must be between the ages of 18 and 99
* Must give consent to participate in the study

Exclusion Criteria:

• Not giving consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 90 years with a diagnosis of diabetes mellitus who gave consent to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Revised Osteoporosis Knowledge Test | 1 day
  The 32-item Revised Osteoporosis Knowledge Test (ROKT; 2012), as reported by Gendler et al. (2015), is a revision of the original 24-item OKT developed by Kim, Horan, & Gendler (1991). This measure was developed to assess the osteoporosis knowledge of adults. Changes were made to update the original OKT to include current recommendations for calcium and vitamin D, exercise requirements, diagnosis and treatment, and a more comprehensive understanding of bone development and osteoporosis risk factors. It contains two subscales (Nutrition and Exercise), which share 14 common items including risk factors and general knowledge. Although the responses offered to participants are multiple choice (e.g., for risk items: more likely, less likely, neutral, don't know), there is only one correct answer for each item. Responses are dichotomously recoded as correct or incorrect.

SECONDARY OUTCOMES:
Osteoporosis Self-Efficacy Scale | 1 day
  The Osteoporosis Self-Efficacy Scale (OSES) utilizes perceived susceptibility and seriousness, perceived barriers and benefits, health motivation, and self-confidence in one's ability to take actions needed to prevent osteoporosis to predict possible occurrence of health behaviors.
Osteoporosis Health Belief Scale | 1 day
  The Osteoporosis Health Belief Scale (OHBS) is a 42-item questionnaire designed to assess susceptibility, seriousness, calcium benefits, calcium barriers, exercise benefits, exercise barriers, and health motivation related to osteoporosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request by the corresponding author.